CLINICAL TRIAL: NCT01411059
Title: Safe and Effective Yoga Prescription of Seniors: Biomechanical Considerations
Brief Title: Yoga Empowers Seniors Study
Acronym: YESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, George Salem, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01AT004869-01 (NIH)
Record Dates: First submitted 2011-07-20; First posted 2011-08-05 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Older Adults
Keywords: yoga biomechanics seniors
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- yoga (Experimental): 32 weeks of yoga training
  Interventions: Behavioral: yoga

INTERVENTIONS:
Behavioral: yoga — yoga classes 2 times per week for 32 weeks
  Other Names: activity intervention

SUMMARY:
This is an Intervention Development Study (IDS) to quantify the physical demands (using biomechanical investigation) of a 2-phase (beginning & intermediate), 32-week yoga program designed for community-dwelling older adults. Additionally, the IDS will explore the adherence and adverse events of participation in the program. Data from the IDS will be used to develop evidenced-based yoga programs, which the investigators postulate will be associated with fewer musculoskeletal side effects compared to non-evidence based yoga programs. The investigators also postulate that evidenced-based tailoring of yoga for seniors will enhance adherence and efficacy. The programs developed during this IDS will be tested in an expanded, Phase II, Randomized Controlled Trial.

DETAILED DESCRIPTION:
Yoga is currently being recommended to restore and preserve strength, flexibility, balance, & physical capacity in older adults; however, our clinical trial experiences suggest that without proper evidenced-based prescription, Yoga participation can be ineffective or even injurious for seniors. To address this lack of evidence-based knowledge, the proposed IDS will: 1) quantify the physical demands of a 32-wk Yoga program designed for independent ambulatory seniors; 2) characterize the relations between these demands and participant physical characteristics; 3) examine the adherence, efficacy, & safety of the program; and 4) characterize the relations among reported adverse events, baseline participant characteristics, and Yoga physical demands.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and women volunteers, aged 65 years or older.

Exclusion Criteria:

* Safety exclusions:

  --the following safety exclusions are adopted in order to decrease potential *cardiovascular
  * musculoskeletal
  * neurological risks to the participants:
* active angina
* uncontrolled hypertension (SBP greater than 160 or DBP greater than 90)
* high resting pulse or respiratory rate (HR >90 or RR>24 after 5 minutes seated)
* unstable asthma or exacerbated COPD
* cervical spine instability or other significant neck injury
* rheumatoid arthritis
* unstable ankle, knee, hip, shoulder, elbow, or wrist joints
* hemiparesis or paraparesis
* movement disorders (e.g. Parkinson's disease), peripheral neuropathies, stroke with residual deficits, severe vision or hearing problems
* walker or wheelchair use
* insufficient hearing to permit safety in a yoga group setting
* not able to attend in-person classes
* has not had check-up by regular provider within 12 months (if not taking any prescription medications) or in the past 6 months (if any regular medicines taken); cannot pass specific movement safety tests (tests described in section on screening visits, below)
* Feasibility/adherence exclusions:

  1. unable to understand their commitment to the project, (laboratory visits & regular program participation)
  2. cognitive limitations significant enough to preclude informed consent or to raise concerns about participation safety

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
peak joint moments | difference from baseline to 16 wk
  These are the torques produced by the muscles during performance of the yoga poses
peak joint moments | difference from 16 wk to 32 wk
  These are the torques produced by the muscles during performance of the yoga poses

SECONDARY OUTCOMES:
time to stand and sit from a chair 5 times | baseline, 16 and 32 weeks
  In the 5-Repetition Chair Stand Test, we record the time it takes for a participant to repeatedly stand and sit on a chair 5 times.
number of heel-rise repetitions | baseline, 16 and 32 weeks
  The Heel-Rise Test is a measure of plantar-flexion endurance. Here, we record the number of full range-of-motion, heel-rise repetitions the participants can complete before fatigue.
Time to complete Up & Go test | baseline, 16 and 32 weeks
  In the Up & Go Test, a measure of mobility, we record the number of seconds it takes to rise from a chair, walk 8 feet, return and sit in the chair.
Number of marching steps completed within 2 minutes | baseline, 16 and 32 weeks
  In the 2-Minute Step Test, a measure stepping endurance, we record the number of complete marching steps the participant can perform within a 2-minute period
Distance participant can reach forward from a sitting position | baseline, 16 and 32 weeks
  The sit and reach test measures overall sagittal-plane flexibility. The participant is asked to reach as far as possible toward their dominant limb while remaining seated.
Distance between fingers of opposing hands as participant attempts to touch fingers while reaching posteriorly. | baseline, 16 and 32 weeks
  The Back Scratch Test measures upper extremity flexibility. Here the distance between finger-tips is recorded as the participant reaches posteriorly and attempts to touch opposing hands.
Maximum passive wrist flexion, extension, radial-deviation, and ulnar-deviation, range of motion (in degrees). | baseline, 16 and 32 weeks
  These tests measure the range of motion of the wrist in the sagittal and frontal planes.
Maximum height participant can reach while standing | baseline, 16 and 32 weeks
  Here we quantify the maximum vertical height participants can reach while standing.
Maximum distance participant can reach forward while standing | baseline, 16 and 32 weeks
  THe Maximum Forward Reach test is a measure of strength and flexibility. Here we record the maximum distance the participant can reach forward while standing.
stride length during walking | baseline, 16 and 32 weeks
  Here we quantify the stride length of participants during walking at a self-selected pace.
Maximum joint angle | baseline, 16 and 32 weeks
  Here we quantify the maximum joint angles of the ankle, knee, hip, trunk, shoulder, elbow, and wrist during performance of the yoga poses.
Sway distance of the center of pressure | baseline, 16 and 32 weeks
  Here we quantify the movement of the center of pressure as participants stand as still as possible
Electromyographic activity of muscles | baseline, 16 and 32 weeks
  Here we record the electromyographic activity of the Anterior Deltoid, Triceps surae, Obliques, Rectus Abdominus, Erector Spinae, Gluteus Maximus, Lateral Hamstrings, Vastus Lateralis, Gastrocnemius, and Gluteus Medius, muscles during performance of the yoga poses.
SF-36 score | baseline and 36 weeks
  Health related quality of life and mood will be assessed with the RAND Short Form-36 (Hays, 1993). The SF-36 includes sub-scales that measure: 1) health-related limitations in physical function; 2) health-related limitations in role and in social function; 3) emotional function (including positive and negative mood states); 4) pain.

CONTACTS AND LOCATIONS:
Overall Officials: george salem, phd, Principal Investigator — University of Southern California
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Wang MY, Yu SS, Hashish R, Samarawickrame SD, Kazadi L, Greendale GA, Salem G. The biomechanical demands of standing yoga poses in seniors: The Yoga empowers seniors study (YESS). BMC Complement Altern Med. 2013 Jan 9;13:8. doi: 10.1186/1472-6882-13-8. PMID 23302513